CLINICAL TRIAL: NCT00326703
Title: Investigation to Determine the Effects of Aircraft Cabin Altitudes on Passenger Comfort and Discomfort
Brief Title: Effects of Aircraft Cabin Altitude on Passenger Comfort and Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Boeing Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Boeing001
Record Dates: First submitted 2006-05-15; First posted 2006-05-17 (Estimated); Last update posted 2006-10-17 (Estimated); Status verified 2006-05

CONDITIONS: Acute Mountain Sickness
Keywords: hypoxia; hypobaric; altitude
MeSH Terms: conditions — Altitude Sickness; Hypoxia

INTERVENTIONS:
Procedure: Hypobaric hypoxia

SUMMARY:
Commercial aircraft passengers are exposed to atmospheric pressures ranging from the pressure found at ground level to that encountered in the external environment at 8,000 feet. There is some evidence in the medical literature that symptoms of acute mountain sickness can result from ascent to altitudes of 6,300 to 10,000 feet by unacclimated persons during the first few days following ascent, probably due to the hypoxia that results from breathing air at the reduced ambient pressures at altitude. The logical hypothesis that follows is that exposure to 8,000 feet could cause hypoxia sufficient to adversely affect the comfort and well being of some commercial aircraft passengers on prolonged flights. There is insufficient data in the literature to validate this hypothesis.

Exercise at sea level and at altitude reduces arterial oxygen levels. The logical hypothesis that follows is that the combination of moderate exercise and exposure to altitude could cause hypoxia sufficiently severe to adversely affect the comfort and well being of some people and that the combined effect of exercise and altitude on comfort and well being is greater than the effect of exercise or altitude alone. Again, there is insufficient evidence in the literature to substantiate this possibility.

The purpose of this investigation is to test these hypotheses.

DETAILED DESCRIPTION:
Altitude affects human health and well being through its effect on tissue oxygenation by altering the partial pressure of oxygen in the gas that enters the lungs. The partial pressure of any component of a mixed gas is equal to the total pressure of the gas multiplied by the fraction of the gas that is made up by the component--approximately 78% for nitrogen and 21% for oxygen in air at all altitudes. As altitude increases, total air pressure decreases and consequently, the partial pressures of all component gases, including oxygen, decrease. As air is inhaled, it becomes saturated with water vapor from body tissues, further reducing its partial pressure of oxygen. Tissue oxygenation, measured in terms of partial pressure of oxygen in arterial blood (paO2), is directly related to the partial pressure of oxygen in the gas entering the lungs.

The United States Federal Aviation Agency requires that commercial aircraft be designed so that the barometric pressure in the cabin at maximum cruise altitude exceeds that found in the external atmosphere at 8,000 feet (565 mm Hg).1 The scientific basis for this limit is unclear. Although there is a large body of knowledge concerning the effects of altitude on humans, most of it involves healthy young people at altitudes higher than 8,000 feet. An investigation of the effects of altitude on commercial airline passengers performed by McFarland in 1937 found "…older persons up to 72 years of age respond to moderate altitudes, i.e., up to 16,000 feet, without unusual difficulties." However, the same author went on to conclude, "The human factors analysis presented here would suggest that the comfort and well-being of airline passengers would be significantly benefited by as near sea level conditions as possible. In any event, cabin altitudes of 3,000 - 5,000 feet should not be exceeded." 2, 3 In 1986, the Committee on Airliner Cabin Air Quality of the National Research Council (NRC) concluded, "Similarly, the decrease in oxygen partial pressure (pO2) that occurs at 8,000 feet is safe for normal people, but possibly hazardous for patients with COPD." 4 In a report published in 2001, the NRC concluded that research into the effect of cabin pressure on susceptible persons should be given high priority.5

Acute Mountain Sickness (AMS), a syndrome characterized by headache, anorexia, nausea, vomiting, lassitude and sleep disturbance, the onset of which closely follows ascent to altitude6 has been reported in 12 to 42% of visitors to altitudes ranging between 6,300 and 10,000 feet in the mountains of Colorado.7-12 The time course of these symptoms was not reported in sufficient detail to allow characterization of their onset during the first several hours after arrival at altitude.

Hypoxia-related medical problems during flight are rare..13-18 However, an unpublished statistical model 19 predicts that at 8,000 feet a substantial proportion of persons whose ages are similar to those of commercial aircraft passengers will experience paO2s below the levels at which use of supplemental oxygen is recommended by various medical authorities.20-24 If the recommendations for use of supplemental oxygen are valid,25, 26 it is possible that exposure to these levels of hypoxia for up to 20 hours (the maximum anticipated duration of commercial aircraft flight segments) could adversely affect the comfort and well being of passengers.

Physical exercise has been demonstrated to reduce blood oxygenation in persons with normal and abnormal pulmonary health.27-29 Some members of the aircraft crew perform moderate levels of work as part of their job30-34, and exercise is recommended by some to alleviate the discomfort experienced as a result of the prolonged inactivity encountered in flight. It is unknown if moderate exercise has a beneficial or deleterious effect on the comfort and well being of persons at altitude.

The terms "comfort" and "well being" are commonly used but imprecisely defined. "Comfort" has been defined as the "... circumstance under which one is able to concentrate fully on selected tasks. No attention is given to the maintaining of well being." 35 "Well being" is defined as "The state of being healthy, happy, or prosperous." 36 This investigation will measure the single concept of "comfort and well being" by using the following factors of the Environmental Symptoms Questionnaire IV:

Factor 1, Cerebral Acute Mountain Sickness; Factor 2, Respiratory Acute Mountain Sickness; and Factor 5, Distress.37

Low scores indicate a greater degree of comfort and well being than do high scores.

Mild hypoxia has been reported to cause asymptomatic changes in oxygen saturation, heart rate, blood pressure, visual function, short term memory, and fine motor coordination.38-41 Unpublished studies have found asymptomatic disorders of control of the pupillary muscles, possibly due to an imbalance between sympathetic and parasympathetic nervous control.42

7. STUDY PLAN AND SCHEDULE

7.1 Study environment

Because of the size of the altitude chamber, multiple "runs" will be required at each altitude to evaluate the required number of test subjects. A "run" will consist of appropriate test subject orientation, screening to exclude persons with temporarily disqualifying health conditions (see Section 7.6.5), entry into the chamber, depressurization to the selected altitude, maintenance of that pressure for a period of time not to exceed 20 hours during which outcome data will be collected and recorded, followed by repressurization to sea level, final data collection and recording, and dismissal. A follow up telephone interview will be conducted 5 to 7 days after the chamber run is completed (Attachment 6). The same test subjects will not be used at multiple altitudes.

During the runs, test subjects will be seated in commercial aircraft seats and allowed to sleep, eat, or walk about as they desire within the physical constraints of the altitude chamber. Aircraft-type entertainment (magazines, books, videotapes) will be provided. Food service and restroom facilities will be available in the chamber. Five test subjects will be randomly selected to exercise on a treadmill ergometer at 3 mph for 10 minutes once an hour for 9 hours to simulate create a the metabolic workload of 2500 to 3300 kcal.

Test subjects and in-chamber test personnel will be blinded to the altitude profile of the run. For test altitudes equal to ground level, brief depressurization and repressurization will be carried out to simulate the noise and pressure changes of a run at higher altitudes.

The following environmental parameters will be maintained within the specified limits for each run:

Pressure: Ground level Ambient +/- 2 mm Hg 2000' 707 mm Hg +/- 2 mm Hg 4000' 656 mm Hg +/- 2 mm Hg 6000' 609 mm Hg +/- 2 mm Hg 7000' 586 mm Hg +/- 2 mm Hg 8000' 564 mm Hg +/- 2 mm Hg

The low frequency with which medical emergencies are reported among airline passengers and visitors to mountain resorts suggests that exposure to altitudes are safe. Therefore, asymptomatic effects of altitude on physiologic parameters are not, a priori, considered sufficiently severe to warrant consideration of design change, and are not included in the altitude selection logic described in paragraph 7.3. Physiologic variables will be measured, however, to demonstrate whether or not the hypoxia encountered during the test runs is sufficiently severe to have any effect on the test subjects.

7.2.1 The following outcomes are of primary interest:

Prevalence and severity of the following symptoms: Measured by:

Fainting Observation Shortness of breath Questionnaire Chest Pain Questionnaire Nausea Questionnaire Headache Questionnaire Malaise Questionnaire Short term memory dysfunction Questionnaire Fatigue Questionnaire Fine Motor Coordination Questionnaire

Physiologic/performance measures Measured by:

Heart Rate Pulse oximeter Arterial oxygen saturation Pulse oximeter Visual acuity Snellen eye chart Color perception FM 100 Hue Short term memory Kentucky Comprehensive Listening Test Fine Motor Coordination Purdue Pegboard

7.2.2 Outcomes of secondary interest are:

Prevalence and severity of the following symptoms: Measured by:

Lightheadedness Questionnaire Dizziness Questionnaire Faintness Questionnaire Flushed Questionnaire Chills Questionnaire Sweaty Questionnaire Shivering Questionnaire Tingling Questionnaire Numbness Questionnaire Ear blockage Questionnaire Blurred vision Questionnaire Tunnel vision Questionnaire Sleepiness Questionnaire Nervousness Questionnaire Irritability Questionnaire Restlessness Questionnaire Depression Questionnaire Happiness Questionnaire Combativeness/aggressiveness Questionnaire

An enhanced Environmental Symptoms Questionnaire (ESQ IV) will be used to ascertain symptom outcomes37. The enhancement consists of additional questions that elicit information concerning the test subjects' perceptions of the chamber environment, recent food and drink intake, and level of activity. It will be distributed prior to depressurization and periodically throughout the run to ascertain the prevalence of symptoms, and an in-chamber attendant will perform the physiologic and performance testing at selected times throughout the run.

7.5 Location of study:

The Center for Aerospace and Hyperbaric Medicine Oklahoma State University Center for Health Sciences 801 East 91st Tulsa Oklahoma 74132

7.6 Test subjects:

Test subjects will be recruited from Tulsa and the surrounding areas. Test subjects will be given $18.00 per hour by Oklahoma State University as compensation for their participation in this study.

The following test subject selection criteria will be used to select a total of 216 test subjects, 108 of whom will be randomly assigned in age strata to 0 and 8,000'. Should the null hypothesis be rejected, 108 test subjects will be recruited for similar assignment to each test altitude. This will be repeated until the altitude selection algorithm has been completed.

7.6.1. Age Distribution:52

Age Sedentary Proportion Sedentary (63 subjects) Exercising Proportion Exercising (45 subjects) Total # < 30 11% 7 28% 13 20 30 - 39.9 17% 10 42% 19 29 40 - 49.9 25% 16 24% 11 27 50 - 59.9 25% 16 6% 2 18 60+ 22% 14 - - 14 Total 100% 63 100% 45 108

7.6.2. Gender Distribution for test subjects will be approximately 50% male and 50% female.

7.6.3. Have flown on commercial flights during past 60 months, but not for 3 or more hours in past 1 month.

7.6.4. Have not been above 4,000' in past 1 month.

7.6.5. Medical History

Do not have a history of:

Lung disease requiring medication or oxygen therapy at ground level Any of the following conditions at AMA Class 3 or worse Chronic Obstructive Lung Disease Chronic bronchitis/emphysema Asthma Restrictive Lung Diseases Any of the following cardiac conditions at AMA Class 3 or worse Coronary Artery Disease Arrhythmia Congestive Heart Failure Cerebrovascular disease Cerebrovascular accident (stroke) Lower Extremity Deep Vein Thrombosis Diabetes mellitus, poorly controlled (change in medication doseage/ frequency in past month) Seizure within past 6 months. Claustrophobia that would impair chamber participation Musculoskeletal disorder that impairs self care and self locomotion. Current anemia of any cause Sickle Cell Anemia Sickle Cell Trait Other conditions, which, in the opinion of the Principal Investigator, might result in excessive risk upon exposure to a hypobaric environment.

Shall not, at the time of the test:

have a contagious disease (including upper respiratory illness) be pregnant be within 4 weeks of a major surgical procedure. have dental abscesses have been scuba diving within 24 hours of test have donated blood within 24 hours of test be under the influence of drugs or alcohol

Health status to be ascertained by questionnaire and interview before each chamber run. Applicants who successfully complete the health questionnaire will undergo a phyical examination by a qualified physician focusing on cardiovascular and pulmonary status before final determination of eligibility will be made. Normal cardiovascular and pulmonary examinations will be required for the applicant to be eligible for inclusion in the study. Test subjects over 40 years of age who will be exercising at altitude will be required to demonstrate their ability to exercise safely to 4.0 METS in a graded exercise tolerance test to be performed before the day of the altitude chamber run.

A "PreRun" questionnaire will be administered the morning of the run before test subjects enter the altitude chamber to determine if the test subjects have developed any disqualifying conditions since undergoing the physician review. All PreRun questionnaires will be reviewed by a Physician Investigator.

7.6.6. Do not have special dietary needs.

7.6.7. Can read and speak English.

All questionnaires, routine and emergency instructions will be given in English. There are no racial or ethnic exclusionary criteria.

7.6.8. Body Size: Body mass index less than 35 and Height less than 74".

The size of the commercial aircraft seats and the altitude chamber interior necessitate a size limitation for the safety and comfort of participants.

7.6.9 Informed Consent: No applicant who has not voluntarily given informed consent to participate will be allowed to participate in this study. Applicants will be given a draft copy of the Informed Consent form to review when they are informed of the dates of orientation sessions. The Informed Consent will be explained in detail during the orientation, and all test subjects' questions concerning it and their participation in the study will be explained. Only Physician and Scientific Researchers will obtain informed consent from the candidates. All signed Informed Consent forms will be retained in accordance with the Boeing Safety, Health, and Environmental Master Records Retention Schedule.

8. STUDY EQUIPMENT AND PROTOCOLS

8.2 Protocols:

The detailed timeline of each run is given in Attachment 4. No test equipment will be attached to the test subjects for the duration of the run. However, the detector of the pulse oximeter will be intermittently clipped to each test subject's finger to measure blood oxygenation. For each measurement, the detector will be attached for approximately 1 minute. Throughout the test protocol from hour 2.5 till hour 14, the test subjects will be provided with video entertainment and magazines, as they would have on a flight. Videos will be stopped during survey times. The test subjects will be asked to bring with them those items they normally take on a flight (books, work, etc.) and to wear clothing that they would wear for a 20 hour flight.

At least one member of the team of investigators will be present in the altitude chamber at all times during the test runs to conduct the testing and to monitor the condition of the test subjects.

Test subjects will be removed from the altitude chamber for the following reasons:

1. Test subject request
2. Any of the following medical conditions:

   Loss of consciousness Chest pain that persists more than 5 minutes Shortness of breath not relieved by reassurance Repeated vomiting
3. Any other condition, which, in the judgment of the in-chamber observer or physician, warrants removal for the safety of the test subjects.

Once a test subject leaves the chamber, he/she will not be allowed to return.

Altitude chamber runs will be scheduled to begin (Hour 0) at 9:00 am. Test subjects will complete testing at approximately 6:30 am the following morning

The duration of the runs may be decreased if it is found that symptom prevalence and severity plateau before 20 hours. This will be determined after all the sea level and 8,000' runs have been completed.

8.3 Research Methodology, Sampling and Data Analysis

8.3.1 Research Methodology

To determine the effects of moderate altitude exposure on comfort and well being, 108 test subjects will be exposed to 8,000 foot-equivalent barometric pressure in an altitude chamber for 20 hours and their responses to symptom survey questions will be compared to responses from 100 test subjects exposed to ambient (ground) pressure for 20 hours in the same chamber.

The study will employ a Split-Split Plot Factorial design. The chamber runs are the whole-plot units and the altitude (0', 8,000' and any intermediate altitudes) is the whole-plot factor, a test subject is the split-plot unit with exercise as the split-plot factor [Ex (exercise) vs Sed (sedentary)], and the repeated measurements on each test subject represent the split-split unit with exposure time as the split-split plot factor. So under this design the appropriate experimental unit for testing altitude differences is a chamber run. The repeated measures in this study include the responses to the symptom items on the questionnaires, which will be administered x times over the 20-hour time period, and the measurements of PaO2, heart rate, etc., which will also be taken repeatedly over the time of the study.

8.3.2 Sampling

Two hundred sixteen test subjects will serve in the study-approximately half will be female and approximately half will be male. The age distribution breakdown is given in the table below (note that for a given age range, approximately half of the test subjects will be male and approximately half will be female). First, 216 test subjects will be selected that fit the distribution given below. Then test subjects of a given gender within a given age range will be randomly assigned to one of four conditions (0' Condition Ex; 0' Condition Sed; 8,000' Condition Ex; and 8,000' Condition Sed). See Attachment 8 for sample size considerations.

0' Condition 8,000' Condition Age # of Subj Ex M/F Sed M/F Ex M/F Sed M/F Ex M/F Sed M/F < 30 40 13/13 7/7 6/7 4/3 7/6 3/4 30 - 39.9 58 19/19 10/10 10/9 5/5 9/10 5/5 40 - 49.9 54 11/11 16/16 5/6 8/8 6/5 8/8 50 - 59.9 36 2/2 16/16 1/1 8/8 1/1 8/8 60+ 28 - 14/14 - 7/7 - 7/7 Total 216 45/45 63/63 22/23 32/31 22/23 31/32

8.3.3 Data Collection and Confidentiality

Survey and telephone interview forms used for collection of test subject responses are shown in Attachment 5. Data recording forms are shown in Attachment 6. The test subjects will be identified on the survey forms by Test Subject Number alone. Data will be entered into an electronic spread sheet using the Test Subject Number as identifier. To insure data integrity, a spreadsheet linking Test Subject Number to name of test subject will be available to the investigators. Spread sheets will reside on file servers protected by password security access. When not in use, survey forms, telephone interview forms, and laptops will be stored in locked cabinets. Paper records will be retained by The Boeing Company and destroyed after 10 years. Electronic data will be stored in password protected computers, or in similarly protected electronic format, indefinitely.

In preparation for data analysis, test subject responses and demographic information will be merged using Test Subject Number, but names will not be included. Only grouped results will be published. Nothing will be published in a form in which the test subject from which the information arose can be identified.

8.3.4 Data Analysis

The symptom data will be analyzed for significant differences between the treatments by first calculating AMS-R, AMS-C and AMS-D from the EQS questions. We will carry out the appropriate Analysis of Variance (ANOVA) for the split-split plot factorial design to look at differences due to altitude and main effects due to activity (Ex vs Sed) and interaction effects between altitude and exercise. This ANOVA will also analyze the within test subject scores to determine if symptom reporting changes over time. Second, the symptoms data will be recoded to "no symptom=0" (0 response on the symptom scale) and "symptom=1" (a 1-6 response on the symptom scale). These data will be analyzed for main effects and interaction effects between altitude and exercise.

The other dependent measures (SaO2, heart rate, etc.) will be analyzed using the appropriate ANOVA for the split-split plot factorial design. These data will also be analyzed for main effects (altitude and activity) and for changes over time, and for the altitude/activity interaction.

ELIGIBILITY:
Inclusion Criteria: age 21 - 75

Exclusion Criteria:Height greater than 6'2", BMI greater than 45. Specified acute or chronic medical conditions -

-

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2002-10; Study Completion 2003-04

PRIMARY OUTCOMES:
ESQ IV factor scores measured at 2 hour intervals
Oxygen Saturation measured at 2 hour intervals

CONTACTS AND LOCATIONS:
Overall Officials: James M Muhm, MD, MPH, Principal Investigator — The Boeing Company

REFERENCES:
- [Derived] Muhm JM, Rock PB, McMullin DL, Jones SP, Lu IL, Eilers KD, Space DR, McMullen A. Effect of aircraft-cabin altitude on passenger discomfort. N Engl J Med. 2007 Jul 5;357(1):18-27. doi: 10.1056/NEJMoa062770. PMID 17611205